CLINICAL TRIAL: NCT03720457
Title: A Phase I Clinical Trial of Human CD19 Targeted T Cells Injection for Subjects With Relapsed and Refractory CD19-positive Diffuse Large B-cell Lymphoma and Follicular Lymphoma
Brief Title: Human CD19 Targeted T Cells Injection(CD19 CAR-T) Therapy for Relapsed and Refractory CD19-positive Lymphoma.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-NHL01; CTR20181354 (Other: National Medical Products Administration)
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: CD19-positive; Diffuse Large B-cell Lymphoma; Follicular Lymphoma
Keywords: CD19; CAR-T; Diffuse Large B-cell Lymphoma; Follicular Lymphoma; Relapsed /Refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human CD19 targeted T Cells Injection (Experimental)
  Interventions: Drug: Human CD19 targeted T Cells Injection

INTERVENTIONS:
Drug: Human CD19 targeted T Cells Injection — Autologous genetically modified anti-CD19 CAR transduced T cells

SUMMARY:
To evaluate the safety and tolerance of human CD19 targeted T Cells injection for the treatment of relapsed and refractory CD19-positive diffuse large B-cell lymphoma and follicular lymphoma. Patients will be given a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by a single infusion of CD19 CAR+ T cells.

DETAILED DESCRIPTION:
Participants with relapsed/refractory CD19-positive Diffuse Large B-cell Lymphoma and Follicular Lymphoma can participate if all eligibility criteria are met.Tests required to determine eligibility include disease assessments, a physical exam, Electrocardiograph, CT/MRI , and blood draws.Participants receive chemotherapy prior to the infusion of CD19 CAR+ T cells. After the infusion, participants will be followed for side effects and effect of CD19 CAR+ T cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects with CD19+ B cell lymphomas who have a limited prognosis (several months to <2 year survival) with currently available therapies will be enrolled.

1. 18 to 70 Years Old, Male and female;
2. Expected survival > 12 weeks;
3. Clinical performance status of ECOG score 0-1;
4. Pathology demonstrated that CD19-positive B-cell non-Hodgkin's lymphoma and who meet one of the following conditions:

   1. Relapsed and refractory CD19-positive Diffuse large B-cell lymphoma and Follicular lymphoma: patients previously received at least first-line and second- line treatment and fail to achieve CR;
   2. Disease recurrence after stem cell transplantation, and at least 1 years after stem cell transplantation.
5. It can establish the venous access required for collection, satisfying hemoglobin ≥ 70 g / L, neutrophils ≥ 1.0 × 10 ^ 9 / L, platelets ≥ 50 × 10 ^ 9 / L. Mononuclear cell collection can be determined by the investigators;
6. At least 1 measurable tumor foci according to the 2014 Lugano treatment response criteria;
7. Liver, kidney and cardiopulmonary functions meet the following requirements:

   1. Serum creatinine ≤ 1.5 × ULN;
   2. Left ventricular ejection fraction >50%, no pericardial effusion and no pleural effusion (ECHO examination);
   3. Baseline oxygen saturation > 92%;
   4. Total bilirubin ≤ 1.5 × ULN;
   5. ALT and AST ≤ 3 × ULN.
8. Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

1. In the first 5 years before screening, there are malignant tumors other than diffuse large B-cell lymphoma and follicular lymphoma, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery，and catheter carcinoma in situ after radical surgery;
2. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood HBV DNA titer higher than the upper limit of detection; hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency Viral (HIV) antibody positive; Positive syphilis test;
3. Any unstable systemic disease including, but not limited to, active infection (except for local infection), unstable angina pectoris, cerebrovascular accident or transient cerebral ischemia (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), severe arrhythmia , liver, kidney or metabolic disease requiring medication;
4. Any other diseases could affect the outcome of this trial;
5. Any affairs could affect the safety of the subjects or outcome of this trial;
6. Pregnant or lactating women, or planned pregnancy during treatment or within 1 year after treatment, or a male subject whose partner plans pregnancy within 1 year of their cell transfusion;
7. Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment;
8. Subjects who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use); And subjects treated with systemic steroids (except inhalation or topical use) within 72h prior to cell transfusion;
9. Received CAR-T treatment or other gene therapies before enrollment;
10. Patients with symptoms of central nervous system or brain metastasis or have received treatment for central nervous system or brain metastasis (radiotherapy, surgery or other treatment) within 3 months before enrollment;
11. Subject suffering disease affects the understanding of informed consent or comply with study protocol;
12. The investigators consider other conditions unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 5.0 | 2 years post infusion

SECONDARY OUTCOMES:
Duration of CAR-positive T cells in circulation | 2 years post infusion
Total number of CAR-positive T cells infiltrated into lymphoma tissue | 2 years post infusion
Overall remission rate including complete response and Partial response defined by the standard response criteria for malignant lymphoma. | 90 days post infusion
Duration of Response after administration | 90 days post infusion
Progress Free Survival after administration | 90 days post infusion
Overall Survival after administration | 90 days post infusion
The immunogenicity of Human CD19 targeted T Cells Injection. (HAMA detection of human anti-mouse antibody) | 2 years post infusion

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - The First Affilicated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Tsao ST, Gu M, Fu C, He F, Li X, Zhang M, Li N, Hu HM. A simple and effective method to purify and activate T cells for successful generation of chimeric antigen receptor T (CAR-T) cells from patients with high monocyte count. J Transl Med. 2022 Dec 19;20(1):608. doi: 10.1186/s12967-022-03833-6. PMID 36536403
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338